CLINICAL TRIAL: NCT05897151
Title: Comparative Study Between Continuous Spinal Anesthesia Versus General Anesthesia in Patients With Sepsis
Brief Title: Continuous Spinal Anesthesia Versus General Anesthesia in Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahmoud Rashad Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Rashad Ahmed, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35987/10/22
Record Dates: First submitted 2023-05-07; First posted 2023-06-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Sepsis; Continuous Spinal Anesthesia; General Anesthesia
MeSH Terms: conditions — Sepsis | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous spinal anesthesia (Experimental): Preservative free 0.5% Hyperbaric bupivacaine (AstraZeneca) 5mg + 25mcg fentanyl for the initial dose will be followed by top up doses of 2.5 mg boluses of 0.5% Hyperbaric bupivacaine every 10 minutes until the desired block height is obtained considering patient hemodynamics. Norepinephrine starting dose 0.01 micg/kg/min will be ready for both groups if needed (main arterial pressure < 70 or main arterial pressure decreased more than 20% of preoperative value). The infusion will be through a wide bore Intravenous line. The dose will be titrated up or down according to the patient hemodynamics.
  Interventions: Drug: Continuous spinal anesthesia
- General anesthesia (Active Comparator): After establishing of ASA monitoring, a wide bore cannula (18Gague) will be inserted. Induction will be done by fentanyl (2 mcg/kg), titrating dose. of propofol according to patient hemodynamic response and atracurium (0.5 mg/kg) to facilitate tracheal intubation maintaining End tidal Co2 between 30-40 mmHg.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: Continuous spinal anesthesia — Preservative free 0.5% Hyperbaric bupivacaine (AstraZeneca) 5mg + 25mcg fentanyl for the initial dose will be followed by top up doses of 2.5 mg boluses of 0.5% Hyperbaric bupivacaine every 10 minutes until the desired block height is obtained considering patient hemodynamics.
  Norepinephrine starting. dose 0.01 micg/kg/min will be ready for both groups if needed (Mean arterial pressure < 70 or Mean arterial pressure decreased more than 20% of preoperative value). The infusion will be through a wide bore Intravenous line. The dose will be titrated up or down according to the patient hemodynamics.
  Arms: Continuous spinal anesthesia
Drug: General anesthesia — After establishing of ASA monitoring, a wide bore cannula (18 G) will be inserted. Induction will be done by fentanyl ( 2 mcg/kg ) , titrating dose of propofol according to patient hemodynamic response and atracurium ( 0.5 mg/kg ) to facilitate tracheal intubation maintaining End tidal Co2 between 30-40 mmHg.
  Arms: General anesthesia

SUMMARY:
The anesthetic efficacy and safety of continuous spinal anesthesia and comparing it with general anesthesia technique in sepsis diagnosed patient.

DETAILED DESCRIPTION:
Hemodynamic instability due to high block largely limits the use of conventional dose spinal anesthesia in high-risk septic patients. Hypotension is more common, and also more hazardous, in septic patients, as they may have decreased physiological reserve and compromised blood supply to various vital organs. A smaller dose of local anesthetic reduces the severity and incidence of hypotension during spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 21 years old
* American Society of Anesthesiologists (III, IV) diagnosed with sepsis (Sequential Organ Failure Assessment (SOFA) score ≥ 7)
* Hemodynamically stable and not on vasopressor due to lower limb pathology candidate for spinal anesthesia to drain source of infection.

Exclusion Criteria:

* Patients with known hypersensitivity to local anesthesia.
* Infection at the site of injection.
* Coagulopathy.
* Septic shock.
* Increase of intracranial pressure.
* Severe deformity of the spinal column.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 28 Days postoperative
  Patients' mortality during the first 28 day after surgery

SECONDARY OUTCOMES:
Changes of Heart Rate | UP to 2 hours postoperative
  Heart Rate: pre induction (base line), just after induction then at
  1min, 5min,10min, 15min, 30min,1 hour after induction, at the end of the surgery and 2 hours postoperative
Changes of Invasive Blood Pressure | UP to 2 hours postoperative
  Invasive Blood Pressure: pre induction, just after induction then at
  1min, 5min,10min ,15min, 30min ,1 hour after induction , at the end of the surgery and 2 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author from one year after study completion.
Supporting Information: Study Protocol
Time Frame: From one year after study completion.
Access Criteria: The data will be available upon reasonable request from the corresponding author